CLINICAL TRIAL: NCT06858761
Title: Health Economic Impact of Robot-assisted Bariatric Surgery vs Conventional Laparoscopy: Prospective Multicenter Randomized Controlled Trial
Brief Title: Health-economic Assessment of Robot-assisted Bariatric Surgery
Acronym: ROBOBAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 69HCL24_0757
Record Dates: First submitted 2025-02-20; First posted 2025-03-05 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Obesity
Keywords: Obesity; Bariatric surgery; Robot
MeSH Terms: conditions — Obesity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Prospective multicenter randomized, controlled in 2 parallel groups, single-blind, superiority trial comparing 2 modalities of bariatric surgery (first-line or revision):
  * Robotic surgical strategy
  * Conventional laparoscopic surgical strategy
Who Masked: Participant
Masking Description: Single-blind study: patient will not be informed of the approach (laparoscopic or robotic) which will be used for their intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot-assisted surgical strategy (Experimental): Primary bariatric surgery (According to the recommendations of the High Authority of Health: patient with a BMI ≥40 kg/m2 and/or BMI ≥35 kg/m2 associated with at least one comorbidity and/or BMI between 30 and 35 kg/m2 and suffering from type 2 diabetes) or revision bariatric surgery (for complications or side effects of a previous surgery), using a robotic approach.
  Interventions: Procedure: Robot-assisted surgical strategy; Other: Visual analog scale; Other: EQ-5D-5L questionnaire; Other: Impact of Weight on Quality of Life (IWQOL) questionnaire
- Conventional laparoscopic surgical strategy (Active Comparator): Primary bariatric surgery (According to the recommendations of the High Authority of Health: patient with a BMI ≥40 kg/m2 and/or BMI ≥35 kg/m2 associated with at least one comorbidity and/or BMI between 30 and 35 kg/m2 and suffering from type 2 diabetes) or revision bariatric surgery (for complications or side effects of a previous surgery), using a conventional laparoscopic approach.
  Interventions: Procedure: Conventional laparoscopic surgical strategy; Other: Visual analog scale; Other: EQ-5D-5L questionnaire; Other: Impact of Weight on Quality of Life (IWQOL) questionnaire

INTERVENTIONS:
Procedure: Robot-assisted surgical strategy — Primary or revision bariatric surgery (for complications or side effects of a previous surgery), using a robotic approach. The robot used will be the Da Vinci X or Xi model (depending on the center) from the company Intuitive Surgical.
  Arms: Robot-assisted surgical strategy
Procedure: Conventional laparoscopic surgical strategy — Primary or revision bariatric surgery (for complications or side effects of a previous surgery), using a conventional laparoscopic approach
  Arms: Conventional laparoscopic surgical strategy
Other: Visual analog scale — All patients will have pain evaluation with visual analog scale
Other: EQ-5D-5L questionnaire — All patients will have quality of life assessment with EQ-5D-5L questionnaire
Other: Impact of Weight on Quality of Life (IWQOL) questionnaire — All patients will have Quality of life assessment with IWQOL questionnaire

SUMMARY:
CONTEXT :

Obesity is a serious disease which affects 17% of the french population. Bariatric and metabolic surgery has demonstrated its efficiency and remains the treatment of reference. Over 40,000 bariatric procedures are performed per year, mainly by laparoscopy ; the robotic approach, historically developed by Intuitive Surgical increases rapidly and accounts for 18% of the procedures in the public system. Whereas the robotic approach has demonstrated its superiority toward laparoscopy for prostatectomies and rectal resections, it still has to be demonstrated for bariatric surgery ; some studies report a decrease rate of complications for complexe procedures and selected patients but the literature remains variable and the benefit of the robot in relation to its high cost must be confirmed.

OBJECTIVES:

To conduct a health-economic assessment (i.e. cost-effectiveness ratio expressed as the additional cost per quality adjusted life-year gained) of the Da Vinci robot in bariatric surgery at 1 year, from the Health Care system point of view.

METHOD :

Randomized (482 patients), controlled, single-blind, multicenter, superiority trial comparing two approaches for primary or revisional bariatric surgery: a group benefiting from a robotic approach and a reference group benefiting from a laparoscopic approach. Data from the trial will be matched via the social security number to the French National Health Insurance Information System (SNDS database) in order to collect care consumption. The quality of life will be assessed using the EuroQol-5 Dimension (EQ5D-5L) questionnaire.

PERSPECTIVES:

This study will have a direct impact on patients care, professional practices and public health policy either by validating the value of the robot in bariatric surgery or conversely, by promoting the laparoscopic approach.

HYPOTHESIS :

Robot-assisted bariatric surgery is more expensive than conventional laparoscopy, but the additional costs associated with the robot are partly offset by a reduction in post-operative complications at 1 year, which should also help to improve patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 18 and 70 years old,
* Female or male patients
* Patient eligible for one of the two situations defined below:

  1. Primary bariatric or metabolic surgery, with a BMI corresponding to one of the 3 following situations, in accordance with the french National Authority for Health (HAS) recommendations published in February 2024:

     * 40 kg/m² OR
     * 35 kg/m² with at least one comorbidity that may improve after surgery (e.g.: high blood pressure, sleep apnea syndrome and other severe respiratory disorders, type 2 diabetes, disabling osteoarticular diseases, steatohepatitis not alcoholic, dyslipidemia, osteoarthritis) OR between 30 and 35 kg/m² with uncontrolled type 2 diabetes
  2. Revision surgery for complication and/or side effects of a previous bariatric surgery
* Patient who has benefited from a pluridisciplinary evaluation (medical, surgical, psychiatric), with a favorable opinion for a bariatric.
* Patient who agrees to be included in the study and who signs the informed consent form,

Exclusion Criteria:

* Presence of a severe and evolutive life threatening pathology, unrelated to obesity,
* Pregnancy or desire to be pregnant during the study,
* Patient not affiliated to a French or European healthcare insurance,
* Patient under supervision or guardianship
* Patient who is unable to give consent,
* Patient who does not understand French
* Patient who has already been included in a trial which has a conflict of interests with the present study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 482 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Incremental cost-effectivEness ratio (ICER) | 1 year after surgery
  Ratio expressed as additional cost per Quality Adjusted Life Year gained (cost/QALY) calculated from:
  * Survival and quality of life data (EQ-5D-5L questionnaire)
  * Cost data (micro-costing) and by individual matching with the French National Health Insurance Information System (SNDS database)

SECONDARY OUTCOMES:
Number, type and severity of intraoperative complications | End of the surgery
  Number, type (medical or surgical) and severity of intraoperative complications (during surgery) for each procedure according to the Dindo-Clavien classification.
Number, type and severity of postoperative complications | 1, 3 and 12 months after surgery
  Number, type (medical or surgical) and severity of complications (within 1 year after surgery) for each procedure according to the Dindo-Clavien classification
Pain assessment | 1 day, 2 days and 1 month after surgery
  Pain will be assessed 1 day, 2 days and 1 month after surgery, according to a visual analogic scale (VAS).
  The VAS measures the intensity of pain on a scale from 0 to 10. 0 representing no pain and at the opposite end, 10 representing extreme pain
Readmission rate | 1, 3 and 12 months after surgery
  Number of patients readmitted within 1 year after surgery.
Reintervention rate | 1, 3 and 12 months after surgery
  Number of patients for whom reintervention was necessary within 1 year after surgery.
Quality of life assessment with EQ-5D-5L questionnaire | Before surgery and at 1, 3, 6 and 12 months after surgery
  This questionnaire is divided into 2 parts:
  A first part with the questions called "EQ-5D descriptive system", representing 5 dimensions: Mobility, Personal autonomy, Current activities, Pain and discomfort, Anxiety and depression. The response is based on 5-point scales (1: no problem; 2: mild problems; 3: moderate problems; 4: severe problems; 5: extreme problems or total incapacity).
  This part is completed by a visual analog scale, called "EQ-5D VAS". It consists of a 20 cm line, graduated from 0 to 100, where the patient must indicate how they evaluate their current state of health, 0 being the worst possible state and 100 the best
Quality of life assessment with IWQOL questionnaire | Before surgery and at 1, 3, 6 and 12 months after surgery
  This questionnaire includes five health concepts: mobility, self-esteem, social life, working conditions and sex life. Five answers will be offered to patients for each item and each answer will be assigned a score ranging from 1 to 5. The most pejorative score is 155.
Duration of surgery | End of the surgery
  Operative time expressed in minutes
Length of hospital stay | at hospital discharge, an average of 3 days +- 2 days
  The Length of stay (in days) is based on the number of days of hospitalization from surgery (day of surgery = D0) until the day of discharge
Readmission rate in High Dependency unit and/or intensive care unit | Within 12 months after surgery
  Number of patients for whom readmission rate in High Dependency unit and/or intensive care unit was necessary within 1 years after surgery.
Cost of the initial hospital stay | at hospital discharge, an average of 3 days +- 2 days
  the cost of the initial surgical stay for each group will be calculated using the micro-costing method
ICER in subgroup of patients with preoperative BMI < 50 versus patients with preoperative BMI > 50 kg/m2 | 12 months after surgery
  Ratio expressed as additional cost per Quality Adjusted Life Year gained (cost/QALY)
ICER in subgroup of patients age > 60 years old versus patients age < 60 years | 12 months after surgery
  Ratio expressed as additional cost per Quality Adjusted Life Year gained (cost/QALY)
ICER in subgroup of patients with primary surgery versus patients with revisional surgery | 12 months after surgery
  Ratio expressed as additional cost per Quality Adjusted Life Year gained (cost/QALY)
ICER in subgroup of patients with restrictive surgery versus patients with malabsorptive surgery | 12 months after surgery
  Ratio expressed as additional cost per Quality Adjusted Life Year gained (cost/QALY)
ICER depending on preoperative risk | 12 months after surgery
  Ratio expressed as additional cost per Quality Adjusted Life Year gained (cost/QALY)
Perform a budgeT impact analysis | 5-year modelling
  Financial consequences of adopting robotic from the perspective of the French public health care system at 5 years

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - Département de chirurgie digestive et endocrinienne Groupe Hospitalier Pellegrin Place Amélie Raba Léon 33076 BORDEAUX, Bordeaux
  - Département de chirurgie digestive CHRU Dijon - Hôpital Le Bocage Bd du Maréchal de Lattre de Tassigny 21000 DIJON, Dijon
  - Digestive Surgery Department CHU Grenoble BP217 - 38043 GRENOBLE Cedex 09, Grenoble
  - Service de Chirurgie Générale et Digestive Grand Hopital de l'Est Francilien Site de Marne La Vallée 2-4 Cours de la Gondoire 77600 JOSSIGNY, Jossigny
  - Service de Chirurgie Générale et Endocrinienne CHU de Lille - Hôpital Claude Huriez 1 rue Michel Polonovski 59000 LILLE, Lille
  - Hospices Civils de Lyon - Hôpital Edouard Herriot Chirurgie Digestive et Bariatrique 5 Place d'Arsonval - 69437 Lyon Cedex 03 - FRANCE, Lyon
  - Département de chirurgie digestive et bariatrique CHU de Nantes - Site Hôtel-Dieu - HME 1 Place Alexis Ricordeau 44000 NANTES, Nantes
  - Département de Chirurgie digestive Hôpital de la Source CHU d'ORLEANS 14 Avenue de l'hôpital 45100 ORLEANS LA SOURCE, Orléans
  - Service de Chirurgie Digestive Hépato-bilio-pancréatique et Transplantation Hépatique Chirurgie Bariatrique, coelioscopique et robotique AP-HP - Hôpital Universitaire La Pitié Salpêtrière 47-83 boulevard de l'hôpital 75013 PARIS, Paris
  - Département de chirurgie digestive, oncologique et bariatrique AP-HP - Hôpital Européen Georges Pompidou 20 rue Leblanc 75015 PARIS, Paris
  - Département de chirurgie digestive, œsogastrique et bariatrique AP-HP - Hôpital Bichat - Claude-Bernard 46 Rue Henri Huchard 75018 PARIS, Paris
  - Département de chirurgie viscérale CHU de Poitiers 2 Rue de la Miletrie - CS 90577 - 86000 POITIERS, Poitiers
  - Clinique Chirurgicale Mutualiste 3 rue le verrier - BP 209 42100 SAINT ETIENNE, Saint-Etienne
  - Département de chirurgie digestive et endocrinienne CHU de Strasbourg - Nouvel Hôpital civil Rez-de-chaussée 1 place de l'hôpital BP 426 67091 STRASBOURG cedex, Strasbourg
  - Service de Chirurgie Digestive Hôpital Rangueil - CHU de Toulouse 1 avenue du Pr Jean Poulhès - TSA 50032 31059 TOULOUSE Cedex 9, Toulouse
  - Département de Chirurgie Viscérale Métabolique et Cancérologique Responsable de l'Unité de Chirurgie Endocrinienne Université de Lorraine CHRU de Nancy - Hôpital Brabois adultes 11 allée du Morvan 54511 VANDOEUVRE LES NANCY, Vandœuvre-lès-Nancy